CLINICAL TRIAL: NCT02904863
Title: Study of 'Vascular Competence' Profile and Endothelial Activation in the Hemolytic Uremic Syndrome in Children and Adults
Acronym: SHU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-03; 2012-A00217-36 (Other: ANSM)
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Hemolytic Uremic Syndrome
MeSH Terms: conditions — Hemolytic-Uremic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with HUS (Experimental)
  Interventions: Biological: Extra blood draw samples

INTERVENTIONS:
Biological: Extra blood draw samples

SUMMARY:
The Hemolytic Uremic Syndrome (HUS) is a rare thrombotic microangiopathy (TMA), affecting both children and adults. HUS is characterized by the abnormal occurrence of diffuse thrombosis in the microcirculation resulting in the occurrence of ischemic events affecting especially the kidneys and is associated with hemolytic anemia. One of the major problems encountered in the management of HUS is the absence of reliable marker of treatment response or relapse; conventional hematological markers being too insensitive to judge therapeutic efficacy or identify early relapse. Data from the literature suggest that the endothelial cell is a major target of this syndrome. Our hypothesis is that an initial micro-endothelial activation plays a critical role in the initiation and / or relapse of the disease.The main objective of this study is to define a "vascular competence" profile in a population of patients with typical or atypical HUS; both in the acute phase and in remission of the disease.

DETAILED DESCRIPTION:
The Hemolytic Uremic Syndrome (HUS) is a rare thrombotic microangiopathy (TMA), affecting both children and adults. HUS is characterized by the abnormal occurrence of diffuse thrombosis in the microcirculation resulting in the occurrence of ischemic events affecting especially the kidneys and is associated with hemolytic anemia.Its prognosis is severe, with a mortality of 1% in children, 10% in adults and the occurrence of renal failure in 50% of cases.In its typical form, HUS occurs in the aftermath of a diarrheic intestinal infection by bacteria which produce a Shiga toxin. In its unusual shape, which affects both children and adults, there are genetic abnormalities alternate way of regulating complement proteins explaining frequent relapses.One of the major problems encountered in the management of HUS is the absence of reliable marker of treatment response or relapse; conventional hematological markers being too insensitive to judge therapeutic efficacy or identify early relapse. Data from the literature suggest that the endothelial cell is a major target of this syndrome. Our hypothesis is that an initial micro-endothelial activation plays a critical role in the initiation and / or relapse of the disease through the sudden release of high molecular weight ultralarge von Willebrand factor (UL-vWHf) and procoagulant endothelial microparticles.The main objective of this study is to define a "vascular competence" profile in a population of patients with typical or atypical HUS; both in the acute phase and in remission of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of typical or atypical HUS in acute phase

Exclusion Criteria:

* Patient with positive serological screening test for infection with the HIV.
* Patients with a history of cancer.
* Patients who have undergone organ transplantation or bone marrow.
* Patient with a vivid picture of autoimmune thrombotic thrombocytopenic purpura

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-02-11 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
number of circulating endothelial cells (CECs) and endothelial progenitor cells (EPCs) | 36 months
number of endothelial progenitor cells (EPCs) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No